CLINICAL TRIAL: NCT06249529
Title: Airway Bypass System - Safety and Feasibility Study A SINGLE-CENTER, PROSPECTIVE, SINGLE ARM STUDY TO EVALUATE THE SAFETY AND FEASIBILITY OF THE AIRWAY BYPASS SYSTEM
Brief Title: Airway Bypass - Safety and Feasibility Study
Acronym: AIRWAY
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zoar Engelman (Industry)
Responsible Party: Sponsor-Investigator, Zoar Engelman, CSO, Deerfield Catalyst
Organization: Deerfield Catalyst (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL2001
Record Dates: First submitted 2023-11-15; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Emphysema or COPD
Keywords: COPD; Emphysema
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental): Patients in the interventional arm will receive implant of one or more airway bypass devices.
  Interventions: Device: Airway Bypass

INTERVENTIONS:
Device: Airway Bypass — Bypass stent(s) are implanted to allow air trapped in the parenchyma to escape

SUMMARY:
The objective of this study is to evaluate its safety and feasibility of the Airway Bypass Stent System in patients with severe emphysema. The study will collect clinical data through 12 months to assess procedural and device safety.

ELIGIBILITY:
Inclusion Criteria:

1. Patient between 50 to 80 years old.
2. High Resolution CT scan indicates severe emphysema.
3. Patient has post- bronchodilator FEV1 less than or equal to 50% of predicted.
4. Total Lung Capacity >100% of predicted.
5. Residual volume ≥225 % of predicted.
6. RV/TLC >0.69
7. Patient has marked dyspnea scoring >2 on mMRC scale of 0-4.
8. Patient has stopped smoking for a minimum of 8 weeks prior to entering the study, as confirmed by COHb ≤2.5%.
9. Patient read, understood, and signed the Informed Consent form.
10. Subject has completed a pulmonary rehab within the last year and/or performs regular physical activity.

Exclusion Criteria:

1. Patient has clinically significant sputum production.
2. Patient has a change in FEV1 >20% post-bronchodilator.
3. Patient has a history of recurrent clinically significant respiratory infection, defined as with more than 3 hospital stays in the past 12 months.
4. Patient has uncontrolled pulmonary hypertension defined by right ventricular pressure >50mmHg and/or evidenced by echocardiogram.
5. Patient has an inability to walk less than 140 meters (150 yards) or greater than 450 meters in 6 minutes.
6. Patient has evidence of any other disease that may compromise survival such as lung cancer, renal failure, any other investigator identified diseases.
7. Patient has an inability to tolerate bronchoscopy under anesthesia.
8. Any contraindication to bronchoscopy procedure, including but not limited to:

   1. Untreatable life-threatening arrhythmias
   2. Inability to adequately oxygenate the patient during the procedure
   3. Acute respiratory failure with hypercapnia
   4. Myocardial infarction within 6 months
   5. Previously diagnosed high-grade tracheal obstruction
   6. Uncorrectable coagulopathy
9. Patient has clinically significant bronchiectasis.
10. Patient has giant bullae >1/3 lung volume.
11. Patient has had previous LVR surgery, lung transplant or lobectomy, or still has ELVR devices or other device to treat COPD in either lung.
12. Patient has been involved in other clinical studies within 30 days prior to this study.
13. Patient is taking >20mg prednisone (or similar steroid) daily.
14. Patient on antiplatelet agent (e.g., clopidogrel) or anticoagulant therapy (e.g., heparin or coumadin) or has not been weaned off prior to procedure.
15. Patient has any other disease that would interfere with completion of study, follow up assessments or that would adversely affect outcomes.
16. A known allergy to nitinol.
17. Patient with uncontrolled diabetes as well as overweight patient (BMI >35 kg/m2).
18. Cancer needing chemotherapy in the past two years.
19. Patient with pleural effusion and/or pneumothorax.
20. Patient with a disease history of asthma, cystic fibrosis, interstitial lung disease (ILD), active tuberculosis.
21. Patient with exacerbation of chronic obstructive pulmonary disease (COPD) within the last year which defined as: An acute event with the need of antibiotic treatment or hospitalization.
22. Subject has severe gas exchange abnormalities as defined by: PaCO2 >55 mmHg, PaO2 <45 mmHg on room air.
23. Patient with acute ischemic heart disease, with proven pulmonary hypertension (SPAP >45 mmHg) in echocardiography and/or need for double platelet aggregation inhibition.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 12 Months
  including but not limited to device-related blood vessel perforation, pneumothorax, COPD exacerbation, device migration, device removal, rehospitalization.

SECONDARY OUTCOMES:
Implant Success | 0 Days
  Device success, defined as the successful creation of the fenestration(s) and successful delivery of the stent(s) at the intended target position(s).
Procedural success | 1 Days
  Procedural success, defined as no occurrence of device-related or procedure-related SAEs during the hospital stay.
CAT | 12 Months
  Improvement of the COPD Assessment Test (CAT) score from baseline.
FEV1 | 12 Months
  Improvement in forced expiratory volume in 1 second (FEV1) from baseline
Residual Volume | 12 Months
  Decrease in the Residual Volume (RV) from baseline
6MWT | 12 Months
  Improvement in the 6-minute walk test from baseline
Dyspnea scale | 12 Months
  Improvement in the mMRC dyspnea scale from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Israeli-Georgian Medical Research Clinic Healthycore, Tbilisi, Georgia